CLINICAL TRIAL: NCT07401641
Title: Effect of Dezocine Versus Nalbuphine Combined With Sufentanil on Postoperative Analgesia, Complications, and Free Flap Survival in Patients Undergoing Oral Cancer Radical Surgery: A Randomized Controlled Clinical Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SYSKY-2025-417-01
Record Dates: First submitted 2026-01-19; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Oral Cancer; Postoperative Pain Management; Free Tissue Flaps; Mouth Neoplasms
Keywords: Dezocine; Nalbuphine; Oral Cancer Surgery; Free Flap Reconstruction; Postoperative Analgesia; Randomized Controlled Trial; Flap Survival
MeSH Terms: conditions — Mouth Neoplasms | interventions — dezocine; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dezocine + Sufentanil (Experimental): Participants in this arm receive postoperative patient-controlled intravenous analgesia (PCIA) with a mixture of Sufentanil (1.0 µg/kg) and Dezocine (0.4 mg/kg), diluted to a total volume of 150 ml with normal saline. The PCIA pump is set with no basal infusion, a bolus dose of 2.5 ml, a lockout interval of 15 minutes, and a maximum hourly limit of 15 ml. This intervention begins at the end of surgery.
  Interventions: Drug: Dezocine and Sufentanil combination
- Nalbuphine + Sufentani (Active Comparator): Participants in this arm receive postoperative patient-controlled intravenous analgesia (PCIA) with a mixture of Sufentanil (1.0 µg/kg) and Nalbuphine (1.0 mg/kg), diluted to a total volume of 150 ml with normal saline. The PCIA pump settings are identical to the experimental group: no basal infusion, a bolus dose of 2.5 ml, a lockout interval of 15 minutes, and a maximum hourly limit of 15 ml. This intervention begins at the end of surgery.
  Interventions: Drug: Nalbuphine and Sufentanil combination

INTERVENTIONS:
Drug: Dezocine and Sufentanil combination — Postoperative patient-controlled intravenous analgesia (PCIA) regimen. The intervention consists of a mixture of two drugs: Sufentanil (at a dose of 1.0 µg per kg of body weight) and Dezocine (at a dose of 0.4 mg per kg). This combination is diluted with normal saline to a total volume of 150 ml and administered via a PCIA pump. The pump is programmed with no background infusion, a patient-controlled bolus of 2.5 ml, a lockout interval of 15 minutes, and a maximum hourly limit of 15 ml. The infusion begins at the end of surgery.
  Arms: Dezocine + Sufentanil
Drug: Nalbuphine and Sufentanil combination — Postoperative patient-controlled intravenous analgesia (PCIA) regimen. The intervention consists of a mixture of two drugs: Sufentanil (at a dose of 1.0 µg per kg of body weight) and Nalbuphine (at a dose of 1.0 mg per kg). This combination is diluted with normal saline to a total volume of 150 ml and administered via a PCIA pump. The pump settings are identical to the comparator regimen: no background infusion, a patient-controlled bolus of 2.5 ml, a lockout interval of 15 minutes, and a maximum hourly limit of 15 ml. The infusion begins at the end of surgery.
  Arms: Nalbuphine + Sufentani

SUMMARY:
Background: Oral cancer radical surgery often requires free flap reconstruction. Postoperative pain is severe, and traditional opioids like sufentanil have side effects and may adversely affect tumor biology. Dezocine and nalbuphine are opioid agonist-antagonists with potentially better safety profiles. Their comparative effects on analgesia, complications, and flap survival in oral cancer surgery are unknown.

Objective: To compare the efficacy of dezocine versus nalbuphine, both combined with sufentanil, for postoperative analgesia, and to evaluate their impact on postoperative complications and free flap survival/function in patients undergoing oral cancer radical surgery with flap reconstruction.

Methods: This is a prospective, randomized, double-blind, controlled trial. Sixty eligible patients (aged 18-70, ASA I-III) will be randomly assigned (1:1) to receive postoperative patient-controlled intravenous analgesia (PCIA) with either Sufentanil + Dezocine or Sufentanil + Nalbuphine. The primary outcome is pain intensity assessed by the Visual Analogue Scale (VAS) at 2, 24, and 48 hours postoperatively. Secondary outcomes include flap survival status, sensory function recovery, incidence of adverse events (e.g., nausea, vomiting), and hospitalization duration.

Potential Impact: This study may identify a superior postoperative analgesic regimen that provides effective pain relief while potentially improving flap outcomes and minimizing side effects for oral cancer patients.

DETAILED DESCRIPTION:
Design: Single-center, prospective, randomized, double-blind, active-controlled, parallel-group trial.

Interventions:

Group D: Sufentanil (1.0 µg/kg) + Dezocine (0.4 mg/kg) diluted to 150ml with normal saline for PCIA (no basal infusion, bolus 2.5 ml, lockout 15 min).

Group N: Sufentanil (1.0 µg/kg) + Nalbuphine (1.0 mg/kg) diluted to 150ml with normal saline for PCIA (parameters identical to Group D).

Standardized general anesthesia protocol for both groups.

Primary Outcome: Postoperative pain scores (VAS, 0-10) at rest at 2, 24, and 48 hours after surgery.

Secondary Outcomes:

Flap survival status (e.g., hematoma, dehiscence, necrosis, infection) on postoperative days 1-7.

Flap sensory function: static/dynamic two-point discrimination and Semmes-Weinstein monofilament test on days 1-7.

Incidence of postoperative adverse events (nausea, vomiting, pruritus, dizziness, sedation).

Postoperative hospital stay duration.

Ramsay sedation scores at 2, 24, and 48 hours.

Intraoperative hemodynamics and blood loss.

Sample Size: 60 patients (30 per group). The calculation is based on a pilot study detecting a difference in 24h VAS scores (1.52 vs 2.35, SD=0.89) with 90% power and α=0.05, accounting for a 20% dropout rate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with oral malignant tumor.
2. Scheduled for oral cancer radical surgery with free flap reconstruction at Sun Yat-sen Memorial Hospital.
3. Age between 18 and 70 years.
4. Sign informed consent.

Exclusion Criteria:

1. Use of analgesic medications within two weeks prior to surgery.
2. History of diabetes, arteriosclerosis, or peripheral vascular disease.
3. Use of hormones, chemotherapy, or immunosuppressants.
4. Severe cardiac, pulmonary, hematological, hepatic, or renal diseases.
5. Known allergy to the study drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | At 2 hours, 24 hours, and 48 hours after surgery.
  Pain intensity assessed at rest using the Visual Analogue Scale (VAS). The VAS is a 100-mm horizontal line where 0 mm represents "no pain" and 100 mm represents "the worst pain imaginable." Patients mark their current pain level on the line.

SECONDARY OUTCOMES:
Incidence of Flap Complications | Daily from postoperative day 1 to day 7.
  The occurrence of complications in the transferred free flap, assessed daily by clinical examination. Complications include hematoma, wound dehiscence, skin necrosis, and infection.
Flap Sensory Recovery - Two-Point Discrimination (2PD) | Daily from postoperative day 1 to day 7.
  Sensory function recovery of the flap assessed using a Disk-Criminator to measure static and dynamic two-point discrimination (2PD). Lower values indicate better sensory discrimination.
Flap Sensory Recovery - Light Touch Threshold | Daily from postoperative day 1 to day 7.
  Sensory function recovery of the flap assessed using Semmes-Weinstein monofilaments. The test determines the minimal force (g/mm²) required for the patient to perceive light touch, with lower values indicating better sensitivity.
Incidence of Postoperative Adverse Events | From the end of surgery until 48 hours postoperatively.
  The frequency of common postoperative adverse effects, including nausea, vomiting, pruritus (itching), dizziness, and somnolence (drowsiness), as recorded in patient charts and through direct questioning.
Ramsay Sedation Score | At 2 hours, 24 hours, and 48 hours after surgery.
  Level of sedation assessed using the Ramsay Sedation Scale (scores 1-6, where 1=anxious/agitated, 2=cooperative/oriented/tranquil, 3=responsive to commands only, 4-6=asleep with varying responses to stimulus).
Postoperative Hospital Stay Duration | From the day of surgery until the day of discharge (assessed up to 30 days).
  The total length of hospitalization (in days) from the day of surgery until the day of discharge, meeting standard discharge criteria.
Intraoperative Hemodynamic Stability | From anesthesia induction until the end of surgery (intraoperative period).
  Measurement of intraoperative stability, including heart rate (beats per minute), blood pressure (mmHg), and peripheral oxygen saturation (SpO2, %). Data points are recorded every 5 minutes.

OTHER OUTCOMES:
Flap Sensory Recovery - Pain Perception | Daily from postoperative day 1 to day 7.
  Sensory function recovery of the flap assessed specifically for pain perception threshold. This is measured using an algesimeter, a device that applies a standardized, gradually increasing mechanical stimulus (e.g., pressure in grams or Newtons) to the flap surface until the patient first reports a sensation of pain. The threshold value (e.g., in grams) is recorded.
Long-term Flap Survival Rate | At 1 month, 6 months, and 1 year after surgery.
  The viability of the free flap assessed clinically. Flap survival is defined as a viable, perfused flap without the need for emergency reoperation due to total necrosis. The outcome is reported as the percentage of patients with a fully surviving flap at each follow-up time point.
One-year Disease-free Survival | At 1 year after surgery.
  The proportion of patients alive without evidence of cancer recurrence (local, regional, or distant) at 1 year after surgery.
Flap Sensory Recovery - Temperature Sensation | Daily from postoperative day 1 to day 7.
  Sensory function recovery of the flap assessed specifically for temperature discrimination. This is measured using the Thissen temperature sensitivity test or similar calibrated thermodes. The test evaluates the ability to distinguish between warm and cold stimuli applied to the flap surface, typically reported as correct identification rates or threshold temperature differences
Flap Contour and Aesthetic Outcome | At 1 month, 6 months, and 1 year after surgery.
  The aesthetic and contour outcome of the reconstructed site is assessed by a surgeon using a standardized visual analog scale (VAS). The assessor rates overall appearance, symmetry, and contour integration with surrounding tissues on a scale from 0 (very poor) to 10 (excellent). The mean VAS score at each time point will be reported.
Oromandibular Functional Recovery | At 1 month, 6 months, and 1 year after surgery.
  Functional recovery related to the flap reconstruction is assessed using a patient-reported outcome measure (PROM) focusing on speech and swallowing.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Sun Yat-sen Memorial Hospital, Sun Yat-sen Universit, Guangzhou, Guangdong, China